CLINICAL TRIAL: NCT03194841
Title: Heart Failure Self-care With the Aid of a Smartphone Application
Acronym: HFSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Marva Foster, Principal Investigator, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15.064
Record Dates: First submitted 2017-06-16; First posted 2017-06-21 (Actual); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heart Failure Application (Experimental): A mobile application that allowed for input of physiologic data, qualitative questions about symptoms and education
  Interventions: Other: Heart failure application

INTERVENTIONS:
Other: Heart failure application — A mobile phone application that allowed for input of physiologic data, qualitative question input and education retrieval along with SMS use.

SUMMARY:
The purpose of this study was the development, and testing of a HF application that was used to provide self-care support to HF patients through a smartphone device. The study appraised current available literature on HF to determine best practices for promoting self-care of HF through direct communication with individuals with HF living at home. For the purpose of this study, smart phone communication was utilized. Smart phone applications allow patients to transmit physiological data, such as weight, blood pressure, heart rate, and symptom data to healthcare providers. Using a secure website, a healthcare worker can access the information and contact the patient via the mobile phone when their data is out of normal range. This study was novel in its approach from what is traditionally offered in that it supported patient self-care decisions by promoting symptom monitoring and offered both tactical and situational skills strategies through at the point education.

ELIGIBILITY:
Inclusion Criteria:

* living in a non-nursing home setting
* primary providers of own self-care
* established diagnosis of heart failure
* cognitively intact
* able to speak/write English

Exclusion Criteria:

* not willing to use a smartphone
* not exhibiting acute decompensated heart failure symptoms

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-08-22 (Actual); Primary Completion 2017-01-06 (Actual); Study Completion 2017-01-06 (Actual)

PRIMARY OUTCOMES:
Self-Care of Heart Failure Index (SCHFI) | two weeks
  Measures how well a person monitors their symptoms, adhere to medication/diet and how confident they are in performing self-care.

SECONDARY OUTCOMES:
Heart Failure Somatic Awareness Scale | two weeks
  It determines the extent of distress associated with heart failure symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Sethares, PhD, Study Chair — University of Massachusetts Dartmouth

IPD SHARING:
Plan to Share IPD: No